CLINICAL TRIAL: NCT06334406
Title: Study of Antitumor T Cell Immune Responses in Patients With Bladder Cancer
Brief Title: Antitumor T Cell Responses in Patients With Bladder Cancer
Acronym: immunoBLAD
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 098 DRC 210 ER03 012
Record Dates: First submitted 2024-02-28; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort A: Patients treated with intravesical instillations for non-invasive bladder cancer
  Interventions: Other: Biological samples
- Cohort B: Patients treated with radiotherapy (+/- concurrent chemotherapy) for invasive bladder cancer
  Interventions: Other: Biological samples
- Cohort C: Patients treated with neo-adjuvant chemotherapy for invasive bladder cancer
  Interventions: Other: Biological samples

INTERVENTIONS:
Other: Biological samples — Blood samples will be collected at baseline, after the diagnostic TURBT, and D15 after the end of treatment in each cohort.
  Tumor tissues will be collected at baseline for three patients.

SUMMARY:
The main objective of this study is to evaluate the induction of Th1 anti-TERT responses by treatments in patients with bladder tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing transurethral resection of the bladder (TURBT) for a tumor detected by cystoscopy with a histological diagnosis of a non-infiltrating or muscle-infiltrating tumor
* For muscle-invasive tumors: localized tumors (T2-T3N0M0) or locally advanced (T4N0M0)
* Written informed consent

Exclusion Criteria:

* History of TURBT for a bladder tumor whatever the stage
* Stages N1-3 or M1 on initial assessment
* Patients under immunotherapy, chemotherapy or other immunosuppressive drugs (prednisone or prednisolone ≤ 10 mg/day is allowed)
* History of cancer in the last 3 years other than basal cell carcinoma or non-invasive cervical cancer
* HIV, hepatitis C or B infection
* Patients with any medical or psychiatric condition or disease,
* Patients under guardianship, curatorship or under the protection of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for a bladder cancer
Sampling Method: Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2024-04-02 (Estimated); Primary Completion 2026-04-02 (Estimated); Study Completion 2026-04-02 (Estimated)

PRIMARY OUTCOMES:
Tumor antigen specific T-cell responses | 15 days after the last instillations (cohort A), 15 days after the end of radiotherapy (cohort B), 15 days after the end of neo-adjuvant chemotherapy (cohort C)
  Increase in the post-treatment sample of at least 30% in the level of anti-TERT Th1 lymphocytes in the blood measured by the ELISpot IFN-γ method, compared to the measurement at baseline.

SECONDARY OUTCOMES:
Monitoring of T cells in the blood | 15 days after the last instillations (cohort A), 15 days after the end of radiotherapy (cohort B), 15 days after the end of neo-adjuvant chemotherapy (cohort C)
  Flow cytometry analysis using T cell markers for : activation (ICOS, CD137, OX40), differenciation (CD45RA, CCR7, CD62L, CD95), cytotoxicity (perforin, granzyme B, GNLY, SlamF7) and exhaustion (PD-1, TIM-3, TIGIT, TCF1, CD39)
Monitoring of immune cell death parameters in the blood | 15 days after the last instillations (cohort A), 15 days after the end of radiotherapy (cohort B), 15 days after the end of neo-adjuvant chemotherapy (cohort C)
  ATP and HMGB1 by ELISA test
Monitoring of immune suppressive cells in the blood | 15 days after the last instillations (cohort A), 15 days after the end of radiotherapy (cohort B), 15 days after the end of neo-adjuvant chemotherapy (cohort C)
  Flow cytometry analysis using Treg markers (CD3, CD4, CD25, CD127, Foxp3) and monocytic MDSC (CD14, CD11b, CD33, HLA-DR, and lineage cocktail CD3 CD19 CD56).
Overall survival | Date of death from any cause (within 2 years after the initiation of the treatment)
  Time between the date of diagnosis and the date of death from any cause
Progression-free survival | date of first progression of the disease (within 2 year after the initiation of the treatment)
  Time interval between the date of diagnosis and the date of first progression (local, pelvic, metastatic [extent of the disease by RECIST v1.1]) or death from any cause
Local progression-free survival | date of first local progression of the disease (within 2 year after the initiation of the treatment)
  Time interval between the date of diagnosis and the date of first local progression or death from any cause
Transcriptomic analysis | At baseline
  Expression of genes of the anti-tumor responses in blood and tumor

IPD SHARING:
Plan to Share IPD: Undecided